CLINICAL TRIAL: NCT03528161
Title: Hypersensitive Troponin Performance to Identify Syncope at Risk of Serious Adverse Events in the Short Term
Acronym: TROPOCOPE
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Other Study IDs: RC31/18/0118; 2018-A01278-47 (Other: ID-RCB)
Record Dates: First submitted 2018-05-03; First posted 2018-05-17 (Actual); Last update posted 2018-07-09 (Actual); Status verified 2018-07

CONDITIONS: Syncope
Keywords: hypersensitive troponin; risk of serious adverse events; emergency
MeSH Terms: conditions — Syncope; Emergencies

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Measurement of hypersensitive troponin — Telephone follow-up at one month, 3 months and 6 months by a clinical research technician. Collection of serious adverse events, reports of hospitalization.
  The hypersensitive troponin assay will be recently proposed in a short-term risk stratification score after syncope (30 days), the canadian syncope risk score. If hypersensitive troponin benefits from interesting performances it needs to be evaluated prospectively, as measured only in 47.9% of syncope in this study. Hypersensitive troponin could be a prognostic marker of early serious adverse cardiovascular events in syncope.

SUMMARY:
Syncope, a frequent reason for emergency room visits and hospitalization, is a symptom of three major etiological entities: cardiac causes, vaso-reflex causes and orthostatic hypotension. The etiological diagnosis is often uncertain and the prognostic assessment orients the outcome of the patient. The vast majority of syncope management costs are related to hospitalizations. Hospitalization in the immediate aftermath of emergency care is justified by a short-term prognosis. The current relevance of hospitalizations and the prognostic assessment of syncope is questioned.

DETAILED DESCRIPTION:
The improvement of cardiac troponin assay techniques has increased its sensitivity to detect myocardial ischemic conditions, even at the expense of a loss of specificity. Myocardial infarction type 2 is due to an imbalance between needs and oxygen supply to cardiomyocytes at the time of an increase of the first and / or a decrease of the second and is favored by an underlying cardiovascular field fragile. Syncope, because of the low flow that they imply, can be the cause of a type II myocardial infarction on fragile cardiovascular ground.

The study is prospectively conducted in all patients admitted for syncope to assess the actual diagnostic performance of hypersensitive troponin in the syncope risk stratification. The primary benefit is to identify patients at risk of serious cardiac events in the short term. The secondary benefits expected from the study are a decrease in unjustified hospitalizations of patients admitted to the emergency for syncope and thus a decrease in the cost of care.

The validation of the indication of the troponin assay in the stratification of the risk after a syncope passes by its prospective evaluation in a prognostic study.

ELIGIBILITY:
Inclusion Criteria:

* Patients admitted to the emergency department for syncope as defined by European Society of Cardiology (ESC) recommendations.

Exclusion Criteria:

* Patient under guardianship or safeguard of justice
* Refusal to participate
* Inability to contact the patient again at M1, M3, M6
* Malaise without loss of consciousness (lipothymia)
* Loss of post-traumatic knowledge (after head trauma)
* Loss of consciousness of toxic origin
* Loss of consciousness of confirmed epileptic origin (known epileptic or strongly evocative history with post-critical state)
* Diagnosis performed during the initial emergency assessment of a major adverse cardiovascular event.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Knowing that the number of malaise admitted per year to emergencies is 3972 (2016 data), and 20% are syncope (about 800 syncope per year), recruitment can be done in 12 months.
  248 patients admitted for syncope.
Sampling Method: Non-Probability Sample
Enrollment: 248 (Estimated)
Dates: Start 2018-06-19 (Actual); Primary Completion 2019-12 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
The sensitivity of hypersensitive troponin in predicting a major undesirable cardiovascular adverse event | 30 days
  The sensitivity of hypersensitive troponin in predicting the occurrence within 30 days of a major undesirable cardiovascular adverse event Positive and negative likelihood ratios (defined from sensitivity and specificity) will also be estimated.
  The definition of a major cardiovascular adverse event was chosen based on recommendations published in the Academy of Emergency Medicine (38) and the American College of Emergency Medicine The primary endpoint will be evaluated in all patients within 30 days of the troponin assay, blinded to the outcome of the biological variable.
The specificity of hypersensitive troponin in predicting a major undesirable cardiovascular adverse event | 30 days
  The specificity of hypersensitive troponin in predicting the occurrence within 30 days of a major undesirable cardiovascular adverse event Positive and negative likelihood ratios (defined from sensitivity and specificity) will also be estimated.
  The definition of a major cardiovascular adverse event was chosen based on recommendations published in the Academy of Emergency Medicine (38) and the American College of Emergency Medicine The primary endpoint will be evaluated in all patients within 30 days of the troponin assay, blinded to the outcome of the biological variable.

SECONDARY OUTCOMES:
The positive and negative predictive values of hypersensitive troponin | 6 months
  The positive and negative predictive values of hypersensitive troponin in the prediction of short-term serious events
The hypersensitive troponin performance | 6 months
  The hypersensitive troponin performance (sensitivity) in the prediction of the occurrence of a major adverse cardiovascular event at 3 and 6 months after syncope

CONTACTS AND LOCATIONS:
Overall Officials: Frédéric Balen, MD, Principal Investigator — University Hospital, Toulouse
Locations (1):
- University Hospital Toulouse, Toulouse, France

IPD SHARING:
Plan to Share IPD: No